CLINICAL TRIAL: NCT02660437
Title: Carbon Dioxide Partial Pressure Oscillations During Exercise: Relation to Cerebral Blood Flow Regulation and and to the Prevalence of Cognitive Dysfunction in COPD
Brief Title: pCO2 Oscillations During Exercise: Relation to Cerebral Blood Flow and to Cognitive Dysfunction in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: European Respiratory Society (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Dr. med., Head physician, Schön Klinik Berchtesgadener Land
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RESPIRE2-8465
Record Dates: First submitted 2016-01-08; First posted 2016-01-21 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Carbon dioxide partial pressure (pCO2); Cerebral blood flow (CBF); Cognitive dysfunction; Mild/Moderate Cognitive Impairment (MCI); Pulmonary Rehabilitation (PR); Standardized Mini Mental State Examination (SMMSE); Addenbrooke's Cognitive Examination (ACE-R); Montreal Cognitive Assessment (MoCA); Telephone Interview for Cognitive Status (TICS); Stroop test (Reaction Time)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Effect of PR in MCI-group (Active Comparator): Evaluation of the acute effect of a 3-week Pulmonary Rehabilitation (PR) program in cognitive function of MCI-Group using SMMSE, ACE-R, MoCA, TICS and Stroop test clinical instruments in reference to potential changes in pCO2 oscillation patterns (post-PR). Intervention: Pulmonary Rehabilitation program; 12 sessions of exercise training/breathing techniques.
  Interventions: Other: Pulmonary Rehabilitation program
- Effect of PR in control-group (Placebo Comparator): Evaluation of the acute effect of a 3-week Pulmonary Rehabilitation (PR) program in cognitive function of control-group using SMMSE, ACE-R, MoCA, TICS and Stroop test clinical instruments in reference to potential changes in pCO2 oscillation patterns (post-PR).
  Intervention: Pulmonary Rehabilitation program; 12 sessions of exercise training/breathing techniques.
  Interventions: Other: Pulmonary Rehabilitation program

INTERVENTIONS:
Other: Pulmonary Rehabilitation program — Patients will attend a comprehensive 3-week PR program (12sessions/ 60min·day) including high intensive interval exercise equivalent to 100% of peak work rate (WRpeak) with 30sec work periods interspersed with 30sec rest periods for 30min and light resistance training (3muscle groups/ 4sets each/10repetitions; ~30min).
  Other Names: Exercise intervention

SUMMARY:
Investigators wish to identify a relationship between substantial changes in carbon dioxide partial-pressure (pCO2), which frequently occur during the transitions from rest to exercise (ΔpCO2 >4 millimeters of mercury [mmHg] from baseline), and the prevalence of cognitive dysfunction in COPD. In particular, it is anticipated to investigate the vascular effect of pCO2 oscillations in the regulation of cerebral blood flow (CBF) during exercise and its impact on cognitive function in Chronic Obstructive Pulmonary Disease (COPD). Furthermore, this study aims to examine whether major pCO2 oscillations have prognostic value in cognitive deterioration at 6, 12, and 18-month follow-up. In addition, the acute effect of 3-week pulmonary rehabilitation (PR) on cognitive function will be explored. The evaluation of cognitive function will be performed by the use of Standardized Mini Mental State Examination (SMMSE), Addenbrooke's Cognitive Examination (ACE-R), Montreal Cognitive Assessment (MoCA), and Telephone Interview for Cognitive Status (TICS) assessing several cognitive domains (cognitive scores) whereas Stroop test [color reading interference] will be used for measuring cognitive performance (Reaction-Time).

DETAILED DESCRIPTION:
Cerebral Blood Flow (CBF) regulation is crucial for the adequate oxygen supply to the brain and the sustenance of cerebrovascular reserve capacity. A fundamental physiologic regulator of CBF is the carbon dioxide partial pressure (pCO2), which determines the dilatation or contraction of cerebral vasculature. CBF regulation response has been found to be strongly dependent upon pCO2 but much less so upon changes in arterial oxygen saturation. CBF is highly sensitive to pCO2 changes which cause pronounced-vasodilatation in increased pCO2 (CBF augmentation) or vasoconstriction in decreased pCO2 levels (CBF diminution). During cerebral activation and increased metabolism, cerebral arterioles dilate contributing to increase CBF but this process is often challenged during exercise and has a potential impact on cognitive function. CBF is linked to cognitive function while serum level of Brain Derived Neurotrophic Factor (BDNF) has been shown as a critical driving force behind neural plasticity with a potential utility as a biomarker of cognitive decline.

Investigators assume that major pCO2 oscillations during exercise (ΔpCO2 >4 millimeters of mercury [mmHg] from baseline) as a reflection of the abnormality in ventilatory efficiency/drive, lead to overall and local disturbances of cerebral blood flow (CBF) and thus can be associated to increased prevalence of cognitive dysfunction in patients with Chronic Obstructive Pulmonary Disease (COPD). Moreover, investigators hypothesize that patients with major pCO2 oscillations during exercise may develop worse cognitive impairment in several cognitive domains and greater cognitive decline compared to "isocapnic" patients at 6, 12, and 18-month follow-up. Inpatient PR may benefit cognitive function by improving breathing (diminishing pCO2 oscillations), therefore improving CBF, and by increasing cerebral neural activation through exercise.

With regard to cognitive dysfunction, which is associated to increased all-cause mortality and disability, investigators wish:

(A) to detect a relationship between major pCO2 oscillations during exercise and increased prevalence of cognitive dysfunction in COPD; (B) to investigate the impact of different pCO2 transitory-patterns (1. pCO2: decline/ hypocapnic, 2. steady/ isocapnic, 3. increase/ hypercapnic) on CBF regulation and cognitive function; (C) to examine whether major pCO2 oscillations can be a determinant of greater cognitive deterioration in several cognitive domains at 6, 12, and18-month follow-up and (D) to explore the acute effect of 3-week PR on pCO2 oscillations and CBF in respect to cognitive function in COPD patients with cognitive impairment.

The evaluation of cognitive function will be performed by the use of Standardized Mini Mental State Examination (SMMSE), Addenbrooke's Cognitive Examination (ACE-R), Montreal Cognitive Assessment (MoCA) and Telephone Interview for Cognitive Status (TICS) assessing several cognitive domains (cognitive scores) whereas Stroop test will be used for measuring cognitive performance (Reaction-Time).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Obstructive Pulmonary Disease (COPD) in Global Initiative on Obstructive Lung Disease (GOLD) stages II to IV
* COPD patients with mild to moderate cognitive impairment (MCI-group: n=100) and without cognitive impairment (Control-group: n=60)
* Normotensive (Blood Pressure range: 101-143/62-91 millimeters of mercury [mmHg])

Exclusion Criteria:

* Resting partial pressure of oxygen in arterial blood (paO2) <55 millimeters of mercury [mmHg]
* Resting partial pressure of carbon dioxide in arterial blood (paCO2) >45 millimeters of mercury [mmHg]
* last exacerbation ≤4weeks
* severe cognitive impairment/dementia
* other neuropsychiatric symptoms

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Carbon-dioxide partial pressure oscillations (ΔpCO2, mmHg) | Day 4-21
  Changes in transcutaneous pCO2 (ΔpCO2, mmHg from baseline values) during Cycle-Endurance Test (CET) at 75% of peak Work Rate (WRpeak). The pCO2 oscillations will be transcutaneous monitored and continuously recorded by the use of "SenTec" Digital Monitoring System (pre/post measurements): 1st measurement during a CET prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement during a CET at the end of PR program (post-PR).

SECONDARY OUTCOMES:
Cognitive Dysfunction (yes/no) | Day 1-3
  Screening of Cognitive Dysfunction according to Petersen's criteria:
  1. Consistent memory complaints preferably corroborated by a close-informant.
  2. Objective characterization of specific deficits in memory and/or other cognitive domains, as indicated by a poor performance on MoCA (<26 points), MMSE (<25 points), ACE-R (<88 points) and TICS (<33 points).
  3. Preserved ability to perform activities of daily living (ADLs), or minimal impairment if considering instrumental ADLs.
  4. Normal global cognitive function.
  5. Absence of dementia (Clinical Dementia Rating Scale (CDR ≤1 point)).
Cognitive Impairment (Standardized Mini-Mental State Examination [SMMSE, scores]) | Day 1-21
  Evaluation of Cognitive Impairment (CI) by the use of clinical instrument of the Standardized Mini-Mental State Examination (SMMSE, scores); 1st measurement prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement at the end of PR program (post-PR).
Cognitive Impairment (Addenbrooke's Cognitive Examination [ACE-R]) | Day 1-21
  Evaluation of Cognitive Impairment (CI) by the use of clinical instrument of the Addenbrooke's Cognitive Examination (ACE-R scores); 1st measurement prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement at the end of PR program (post-PR).
Cognitive Impairment (Montreal-Cognitive Assessment [MoCA, scores]) | Day 1-21
  Evaluation of Cognitive Impairment (CI) by the use of clinical instrument of the Montreal-Cognitive Assessment (MoCa scores); 1st measurement prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement at the end of PR program (post-PR).
Cognitive Impairment (Telephone Interview for Cognitive Status [TICS]) | Day 1-21
  Evaluation of Cognitive Impairment (CI) by the use of clinical instrument of the Telephone Interview for Cognitive Status (TICS scores); 1st measurement prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement at the end of PR program (post-PR).
Cognitive Performance (Stroop test [reaction-time, seconds]) | Day 4-21
  Assessment of cognitive performance (Stroop test - reaction-time, seconds) before and immediately after Cycle-Endurance Test (CET) at 75% of WRpeak. Cognitive performance will be measured by the use of Stroop-test (pre/post measurements): 1st measurement during a CET prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement during a CET at the end of PR program (post-PR).
Cerebral Blood Flow Velocity (CBFv, cm/sec) | Day 4-21
  Measurement of Cerebral Blood Flow velocity (CBFv, cm/sec) as surrogate of Cerebral Blood Flow (CBF) before and immediately after Cycle-Endurance Test (CET) at 75% of WRpeak. Cerebral Blood Flow velocity (CBFv) will be measured by the use of transcranial Doppler ultrasonography (pre/post measurements): 1st measurement during a CET prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement during a CET at the end of PR program (post-PR).
Frontal cortex cerebrovascular oxygen saturation (Tissue Oxygen Saturation [TOI, %]) | Day 4-21
  Measurement Tissue Oxygen Saturation (TOI, %) as an index of frontal cortex cerebrovascular oxygen saturation during Cycle-Endurance Test (CET) at 75% of WRpeak. Tissue oxygen saturation (TOI, %) will be continuously measured by the use of Near-Infrared Spectroscopy (NIRS-method; pre/post measurement): 1st measurement during a CET prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement during a CET at the end of PR program (post-PR).
Frontal cortex cerebrovascular oxygen saturation (Changes in Deoxygenated Haemoglobin [ΔHHb, μM/cm]) | Day 4-21
  Measurement of the changes in Deoxygenated Haemoglobin (ΔHHb) in micrometer per centimeter (μM/cm) as an index of frontal cortex cerebrovascular oxygen saturation during Cycle-Endurance Test (CET) at 75% of WRpeak. Changes in Deoxygenated Haemoglobin (ΔHHb, μM/cm) will be continuously measured by the use of Near-Infrared Spectroscopy (NIRS-method; pre/post measurement): 1st measurement during a CET prior to the participation in a 3-week (12 sessions) Pulmonary Rehabilitation program (pre-PR); 2nd measurement during a CET at the end of PR program (post-PR).

OTHER OUTCOMES:
Airflow limitation (Forced Expiratory Pressure in 1 Second [FEV1, %predicted]) | Day 1-4
  Measurement of Forced Expiratory Pressure in 1 Second (FEV1, %predicted).
Exercise capacity (peak Work Rate, [WRpeak watts]) | Day 1-6
  Measurement of exercise capacity by a cardiopulmonary exercise test (CPET) on cycle ergometer using an incremental protocol to the limit of tolerance (peak Work Rate, watts)) for establishing the work rate corresponding to 75% of peak (maximum working capacity) according to the international guidelines.
Blood Gas Analyses (Arterial oxygen partial pressure [PaO2, mmHg]) | Day 1-6
  Measurement of arterial oxygen partial pressure (PaO2, mmHg) in blood samples.
Blood Gas Analyses (Arterial carbon-dioxide partial pressure [PaCO2, mmHg]) | Day 1-6
  Measurement of arterial carbon-dioxide partial pressure (PaCO2, mmHg) in blood samples.
Brain Derived Neurotrophic Factor (BDNF serum levels, ng/mL). | Day 1-8
  Measurement of serum levels of Brain Derived Neurotrophic Factor (BDNF, ng/mL) in blood samples.
Psychological condition/ Psychological data (Hospital Anxiety and Depression Scale [HADS, scores]) | Day 5-8
  Psychological factors will be assessed by the use of the Hospital Anxiety and Depression Scale (HADS).
Psychological condition/ Psychological data (COPD Assessment Test [CAT, scores]) | Day 5-8
  Psychological factors will be assessed by the use of the COPD Assessment Test (CAT).
Psychological condition/ Psychological data (St. George Respiratory Questionnaire [SGRQ, scores]) | Day 5-8
  Psychological factors will be assessed by the use of the St. George Respiratory Questionnaire (SGRQ).
Perception of Dyspnoea (Medical Research Council dyspnoea scale, [MRC scores]) | Day 5-8
  Perception of dyspnoea will be assessed by the use of the Medical Research Council (MRC) dyspnoea scale.

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Prof. med., Study Chair — Schön Klinik Berchtesgadener Land
Locations (1):
- Klinikum Berchtesgadener Land der Schön-Kliniken, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Payne SJ, Mohammad J, Tisdall MM, Tachtsidis I. Effects of arterial blood gas levels on cerebral blood flow and oxygen transport. Biomed Opt Express. 2011 Mar 25;2(4):966-79. doi: 10.1364/BOE.2.000979. PMID 21483617
- [Background] Ogoh S, Tsukamoto H, Hirasawa A, Hasegawa H, Hirose N, Hashimoto T. The effect of changes in cerebral blood flow on cognitive function during exercise. Physiol Rep. 2014 Sep 28;2(9):e12163. doi: 10.14814/phy2.12163. Print 2014 Sep 1. PMID 25263210
- [Background] Shimada H, Makizako H, Doi T, Yoshida D, Tsutsumimoto K, Anan Y, Uemura K, Lee S, Park H, Suzuki T. A large, cross-sectional observational study of serum BDNF, cognitive function, and mild cognitive impairment in the elderly. Front Aging Neurosci. 2014 Apr 15;6:69. doi: 10.3389/fnagi.2014.00069. eCollection 2014. PMID 24782766
- [Background] Ito H, Ibaraki M, Kanno I, Fukuda H, Miura S. Changes in the arterial fraction of human cerebral blood volume during hypercapnia and hypocapnia measured by positron emission tomography. J Cereb Blood Flow Metab. 2005 Jul;25(7):852-7. doi: 10.1038/sj.jcbfm.9600076. PMID 15716851
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol. 1999 Mar;56(3):303-8. doi: 10.1001/archneur.56.3.303. PMID 10190820
- [Background] Van der Elst W, Van Boxtel MP, Van Breukelen GJ, Jolles J. The Stroop color-word test: influence of age, sex, and education; and normative data for a large sample across the adult age range. Assessment. 2006 Mar;13(1):62-79. doi: 10.1177/1073191105283427. PMID 16443719
- [Background] Valdueza JM, Balzer JO, Villringer A, Vogl TJ, Kutter R, Einhaupl KM. Changes in blood flow velocity and diameter of the middle cerebral artery during hyperventilation: assessment with MR and transcranial Doppler sonography. AJNR Am J Neuroradiol. 1997 Nov-Dec;18(10):1929-34. PMID 9403456
- [Background] Vogiatzis I, Louvaris Z, Habazettl H, Andrianopoulos V, Wagner H, Roussos C, Wagner PD, Zakynthinos S. Cerebral cortex oxygen delivery and exercise limitation in patients with COPD. Eur Respir J. 2013 Feb;41(2):295-301. doi: 10.1183/09031936.00016312. Epub 2012 May 3. PMID 22556019